CLINICAL TRIAL: NCT03056846
Title: Probiotics (Lactobacillus Gasseri KS-13, Bifidobacterium Bifidum G9-1, Bifidobacterium Longum MM-2) on Stress-associated Gastrointestinal Function in University Students: a Randomized, Double-blind, Placebo-controlled Clinical Trial
Brief Title: Probiotics on Stress-associated Gastrointestinal Function in University Students
Acronym: SAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Wakunaga Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: IRB201600917
Record Dates: First submitted 2016-08-26; First posted 2017-02-17 (Actual); Last update posted 2019-03-25 (Actual); Status verified 2019-03

CONDITIONS: Healthy
Keywords: probiotic; gastrointestinal; stress; student

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Placebo (Placebo Comparator): Placebo will be taken as a capsule twice daily for 6 weeks by subjects in the group receiving this supplement (group is unknown, double-blinded).
  Interventions: Dietary Supplement: Placebo
- Probiotic Combination (Experimental): A commercially available probiotic mixture of Lactobacillus gasseri, Bifidobacterium bifidum, and Bifidobacterium longum will be taken as a capsule twice daily for 6 weeks by subjects in the group receiving this supplement (group is unknown, double-blinded).
  Interventions: Dietary Supplement: Probiotic Combination
- Bifidobacterium bifidum (Experimental): A commercially available probiotic strain (Bifidobacterium bifidum) will be taken as a capsule twice daily for 6 weeks by subjects in the group receiving this supplement (group is unknown, double-blinded).
  Interventions: Dietary Supplement: Bifidobacterium bifidum
- Bifidobacterium longum (Experimental): A commercially available probiotic strain (Bifidobacterium longum) will be taken as a capsule twice daily for 6 weeks by subjects in the group receiving this supplement (group is unknown, double-blinded).
  Interventions: Dietary Supplement: Bifidobacterium longum

INTERVENTIONS:
Dietary Supplement: Placebo — Placebo will be taken as a capsule twice daily for 6 weeks by subjects in the group receiving this supplement (group is unknown, double-blinded).
  Arms: Placebo
Dietary Supplement: Probiotic Combination — A capsule containing a mixture of Lactobacillus gasseri, Bifidobacterium bifidum, and Bifidobacterium longum (1.5 billion cells per capsule prior to expiration) will be taken twice daily for 6 weeks by subjects in the group receiving this supplement (group is unknown, double-blinded).
  Other Names: Kyo-Dophilus; Lactobacillus gasseri KS-13; Bifidobacterium bifidum G9-1; Bifidobacterium longum MM-2
  Arms: Probiotic Combination
Dietary Supplement: Bifidobacterium bifidum — A capsule containing Bifidobacterium bifidum (1.5 billion cells per capsule prior to expiration) will be taken twice daily for 6 weeks by subjects in the group receiving this supplement (group is unknown, double-blinded).
  Other Names: Kyo-Dophilus; Bifidobacterium bifidum G9-1
  Arms: Bifidobacterium bifidum
Dietary Supplement: Bifidobacterium longum — A capsule containing Bifidobacterium bifidum (1.5 billion cells per capsule prior to expiration) will be taken twice daily for 6 weeks by subjects in the group receiving this supplement (group is unknown, double-blinded). Inactive ingredients include gelatin, potato starch, and silica.
  Other Names: Kyo-Dophilus; Bifidobacterium longum MM-2
  Arms: Bifidobacterium longum

SUMMARY:
The purpose of this research study is to evaluate the effect of a daily supplement of probiotics (Lactobacillus gasseri KS-13, Bifidobacterium bifidum G9-1, Bifidobacterium longum MM-2) on stress-associated gastrointestinal function in university students during the time of semester exams.

DETAILED DESCRIPTION:
In this randomized, double-blind, placebo-controlled study, undergraduate students planning to take a fall final exam will receive a daily probiotic combination, individual probiotic, or placebo for 6 weeks. Questionnaires will assess gastrointestinal symptoms, immune health, stress and stress management, quality of life, diet, adverse events, and compliance. In a subset of subjects, stool samples will be collected at baseline and at week 5 of the intervention (the week before final exams) to characterize microbial communities.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Healthy full-time undergraduate student at the University of Florida
* Willing and able to consume a daily supplement (probiotic or placebo) for the duration of the 6-week study
* Willing and able to complete daily questionnaires online regarding general health and well-being, including stress levels and gastrointestinal symptoms (Note: we will recruit participants who will have Internet access for the duration of the protocol, but understand that, once enrolled, situations may change. If this is the case, paper copies of the online forms will be provided)
* Willing to discontinue any immune-enhancing dietary supplements (e.g., prebiotics and fiber supplements, probiotics, Echinacea, fish oil, vitamin E [>400% of the RDA or >60 mg/day])
* Had a cold/flu within the past year

Exclusion Criteria:

* Currently smoke
* Women who are lactating, know that they are pregnant, or are attempting to get pregnant
* Currently taking any systemic corticosteroids
* Currently being treated for any physician-diagnosed diseases
* Have received chemotherapy or other immune suppressing therapy within the last year

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 634 (Actual)
Dates: Start 2017-09-05 (Actual); Primary Completion 2017-12-21 (Actual); Study Completion 2018-02-05 (Actual)

PRIMARY OUTCOMES:
Change in Gastrointestinal Symptom Response Scale (GSRS) constipation symptom score | Baseline (Week 0) to Final (Week 6)
  Weekly GSRS constipation symptom score in probiotic mixture vs. individual probiotic vs. placebo

SECONDARY OUTCOMES:
Change in diarrhea symptoms, measured by GSRS | Baseline (Week 0) to Final (Week 6)
  Weekly GSRS diarrhea symptom scores in probiotic mixture vs. individual probiotic vs. placebo
Change in abdominal pain symptoms, measured by GSRS | Baseline (Week 0) to Final (Week 6)
  Weekly GSRS abdominal pain symptom scores in probiotic mixture vs. individual probiotic vs. placebo
Change in indigestion symptoms, measured by GSRS | Baseline (Week 0) to Final (Week 6)
  Weekly GSRS indigestion symptom scores in probiotic mixture vs. individual probiotic vs. placebo
Change in reflux symptoms, measured by GSRS | Baseline (Week 0) to Final (Week 6)
  Weekly GSRS reflux symptom scores in probiotic mixture vs. individual probiotic vs. placebo
Weekly average of daily levels of stress | Baseline (Week 0) to Final (Week 6)
  Daily stress (0 = no stress to 10 = severe or extreme stress)
Microbiota studies, measured by 16S rRNA sequence analysis | Baseline (Week 0) and Week 5
  Microbial diversity measured by 16S rRNA sequence analysis
Microbiota studies, qPCR | Baseline (Week 0) and Week 5
  qPCR to quantify changes in bacteria of interest
Immune health, measured by questionnaire data | Baseline (Week 0) to Final (Week 6)
  Proportion of healthy days (i.e., days without cold symptoms with an intensity >6). Daily health questionnaires ask students about non-allergy-related cold symptoms (running/congested nose, stiffness or chills, headache, cough, fatigue, fever, sore throat, achiness, and ear discomfort) and symptom intensity (0=none, 1=mild, 2=moderate, 3=severe)
Immune function, measured by questionnaire data | Baseline (Week 0) to Final (Week 6)
  Symptom intensity score (average sum of symptom intensities)

CONTACTS AND LOCATIONS:
Overall Officials: Bobbi Langkamp-Henken, PhD, RD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States